CLINICAL TRIAL: NCT05346003
Title: Investigation of the Effect of Blended E-Learning Method Given to Nursing Students on Students' Knowledge and Psychomotor Skills on Basic Life Support: A Pilot Study
Brief Title: The Effect of Blended E-Learning Method on Students' Knowledge and Psychomotor Skills on Basic Life Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Aynur KOYUNCU, Principal Investigator, Assist Prof, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TDSP
Record Dates: First submitted 2022-04-04; First posted 2022-04-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Qualified CPR Education
Keywords: blended e-learning; cardiopulmonary resuscitation; nursing; simulation; CPR mockup

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the pre-test, all students will be given a BLS information form, followed by blended e-learning with theory and video in a virtual environment. he BLS knowledge post-test will be administered immediately after class.T-shirts and standard pillows (550 g silicon fiber pillow 50x70 cm size) with a simulation of an adult human size (approximately) sternum, rib and heart drawing (printed as picture) will be given to the intervention group only after the pretest. In the study, the BLS will be simulated for adult patients only. To simulate a half-body human CPR mock-up, a pre-made simulation t-shirt will be fitted on a standard pillow to create a CPR mock-up in a home environment, and after blended e-learning, they will be able to perform CPR iteratively on a T-shirt-clad simulation pillow (TCSP) model. In this way, autonomous learning will be supported. All students will practice CPR in a real simulation model two weeks after the blended e-learning.
  Interventions: Procedure: TCSP
- Control Group (No Intervention): In the pretest, all students will be given a BLS knowledge test, followed by e-learning blended with theory and video in a virtual environment. The BLS knowledge post-test will be administered immediately after class. Two weeks after the blended e-learning, all students will practice CPR in a real simulation model. Psychomotor skills will be recorded in the evaluation form.

INTERVENTIONS:
Procedure: TCSP — In the pre-test, all students will be given a BLS information form, followed by blended e-learning with theory and video in a virtual environment. The BLS knowledge post-test will be administered immediately after class.T-shirts and standard pillows (550 g silicon fiber pillow 50x70 cm size) with a simulation of an adult human size (approximately) sternum, rib and heart drawing (printed as picture) will be given to the intervention group only after the pretest. In the study, the BLS will be simulated for adult patients only. To simulate a half-body human BLS mock-up, a pre-made simulation t-shirt will be fitted on a standard pillow to create a BLS mock-up in a home environment, and after blended e-learning, they will be able to perform BLS iteratively on a T-shirt-clad simulation pillow (TCSP) model. In this way, autonomous learning will be supported. All students will practice BLS in a real simulation model two weeks after the blended e-learning.
  Arms: Intervention Group

SUMMARY:
The fact that Basic Life Support (BLS) training is factor determining survival necessitates the dissemination of BLS training. However, the fact that BLS training increases the workload of trainers and requires cost is one of the most important obstacles to the dissemination of this training. The search for new training methods with high efficiency and low cost continues in BLS training. Global guidelines recommend increasing quality of BLS and autonomous learning on BLS, and also encourage studies to develop methods related to this.

The use of e-training methods in BLS training is reported to be cost-effective as well as reducing the burden of trainers. In studies investigating the effectiveness of e-learning methods in BLS training, simulation models with feedback were used to evaluate psychomotor skills of the training. In this study, it was evaluated that it would be beneficial to apply a blended e-learning method, which includes video demonstrations of theoretical and BLS psychomotor skills, to nursing students in a virtual classroom environment. In evaluation of the psychomotor skills of BLS training, it was thought that a simple simulation model (Tshirt Dressed Simulation Pillow (TDSP)) could be created in home environment by wearing the tshirt with the sternum and heart print on a standard pillow (40 X 60 cm) in the student's home. It is thought that psychomotor skills will be improved with repetitive BLS applications that students will make on this model in the home environment. Two weeks after blended training, the BLS application will be made and evaluated on the real model. This training and assessment method is a new method that will allow the evaluation of BLS knowledge and the development of psychomotor skills with autonomous learning, and the fact that there is no study on this subject in the literature constitutes the original value of this study.

In this study, it is aimed to evaluate effects of the blended e-training method and TDSP model given to nursing students on the cognitive and psychomotor learning outcomes of the students on BLS.

The research is a randomized, controlled pilot study in a quasi-experimental design to be conducted at Hasan Kalyoncu University, Faculty of Health Sciences, Department of Nursing. The study was approved by Hasan Kalyoncu University Health Sciences Non-Interventional Research Ethics Committee. Written permission will be obtained. Before starting the study, the aims and objectives of the research will be explained to the students, information will be given about the blended e-learning method to be applied in the research, what the students should do within the scope of the research and data collection methods. Written and verbal consent will be obtained from the students who volunteered to participate in the study. The population of the research will be students (N=387) studying at Hasan Kalyoncu University, Faculty of Health Sciences, Department of Nursing in the 2021-2022 academic year. Students who have received BLS training for the first time, who have not practiced BLS before, and who voluntarily agree to participate in the study will be included in the study. The number of samples was determined as n=62 by power analysis. Students who accept to participate will be randomly divided into two groups through the computer program. The data collection tool consists of two forms, the form consisting of the introductory information of the students and the evaluation form of BLS knowledge and skills. The answers given to the cognitive questions and psychomotor skills of the nursing students in the study and control groups in the pre-test and post-test will be compared with appropriate statistical methods. A value of P<0.05 will be accepted for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

First time receiving BLS training, Those who have not applied BLS before, Students who accept to participate in the research voluntarily

Exclusion Criteria:

Students who have received BLS training or applied BLS before and who work as health professionals, The students who want to leave at any stage after participating in the research voluntarily

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-05-28 (Actual); Primary Completion 2022-08-28 (Estimated); Study Completion 2022-09-28 (Estimated)

PRIMARY OUTCOMES:
The effect of repeated applications with t-shirt dressed simulation pillow on psychomotor skills | Two weeks after the blended e-learning
  The students in the study group will repeat the BLS application with the TDSP model given to them after the theoretical and video lessons, and the effect of frequent repetitions on psychomotor skills will be evaluated. The psychomotor skill evaluation form created by the researchers by using literature review will be used. For the content validity of this form, the opinions of five expert professionals who are experienced in their field were taken in accordance with the Davis technique.

SECONDARY OUTCOMES:
The effect of blended e-education on BLS knowledge level | Before the blended e-learning and immediately after the blended e-learning
  It will be evaluated how theoretical and video BLS education affects the level of knowledge compared to classical education. For the evaluation of the information, the BLS Information Evaluation Form, which was created according to the literature review, will be used. For the content validity of this form, the opinions of five expert professionals who are experienced in their field were taken in accordance with the Davis technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aziz K, Lee HC, Escobedo MB, Hoover AV, Kamath-Rayne BD, Kapadia VS, Magid DJ, Niermeyer S, Schmolzer GM, Szyld E, Weiner GM, Wyckoff MH, Yamada NK, Zaichkin J. Part 5: Neonatal Resuscitation: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S524-S550. doi: 10.1161/CIR.0000000000000902. Epub 2020 Oct 21. No abstract available. PMID 33081528
- [Background] Castillo J, Gallart A, Rodriguez E, Castillo J, Gomar C. Basic life support and external defibrillation competences after instruction and at 6 months comparing face-to-face and blended training. Randomised trial. Nurse Educ Today. 2018 Jun;65:232-238. doi: 10.1016/j.nedt.2018.03.008. Epub 2018 Mar 24. PMID 29605787
- [Background] Chen YS, Lin JW, Yu HY, Ko WJ, Jerng JS, Chang WT, Chen WJ, Huang SC, Chi NH, Wang CH, Chen LC, Tsai PR, Wang SS, Hwang JJ, Lin FY. Cardiopulmonary resuscitation with assisted extracorporeal life-support versus conventional cardiopulmonary resuscitation in adults with in-hospital cardiac arrest: an observational study and propensity analysis. Lancet. 2008 Aug 16;372(9638):554-61. doi: 10.1016/S0140-6736(08)60958-7. Epub 2008 Jul 4. PMID 18603291
- [Derived] Koyuncu A, Pehlivan K, Yava A, Cetindas K, Karacan HI, Ulasli Z. New method for autonomous learning of BLS psychomotor skills: Pillow mannequin: Randomized controlled study. Nurse Educ Today. 2024 Sep;140:106273. doi: 10.1016/j.nedt.2024.106273. Epub 2024 Jun 5. PMID 38924976
- See also: Related Info — http://www.ahajournals.org/doi/10.1161/CIR.0000000000000918